CLINICAL TRIAL: NCT00005269
Title: Family Blood Pressure Program - GENOA
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric Boerwinkle, Professor - SPH, The University of Texas Health Science Center, Houston
Other Study IDs: 1153; 5U01HL054481-13 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Coronary Artery Disease

SUMMARY:
To localize, identify, and evaluate common polymorphic variation in genes involved in determining interindividual differences in blood pressure (BP) levels and essential hypertension status in three racial groups: African-Americans, Mexican-Americans, and Non-Hispanic Whites. The study consists of a six grant network, which in turn is part of an NHLBI initiative, the Family Blood Pressure Program (FBPP) consisting of four networks.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension, a complex disease involving the interplay of genetic and environmental factors, affects an estimated 50 million Americans and is a major predisposing factor for myocardial infarction, vascular disease, stroke, and renal failure. It has been estimated from segregation analysis and twin studies that approximately 45 percent of the interindividual differences in blood pressure are accounted for by genetic differences. The identification of the genes whose variants contribute to high blood pressure will have far-reaching effects on our understanding of the pathophysiology of the circulation and may suggest new preventive measures and rational therapeutic approaches.

One of the principal advantages of the genetic approach is that it identifies primary molecular defects. As a result, it will be possible to stratify the general hypertensive population into subgroups based on genotype and intermediate phenotype and thereby evaluate preventive strategies and therapeutic approaches in more homogeneous groups. In addition, the identification of hypertensive genes also provides the basis for an understanding of the interactions between genes and environmental factors. It is very likely that particular environmental variables exert their effects only in the presence of certain genotypes.

Until recently, the techniques for dissecting the genetic determinants of high blood pressure were not available or were not developed to an extent that would make the Family Blood Pressure Program initiative feasible. However, several recent advances in technology and analytical methods, together with the rapid construction of genetic maps, have substantially improved the chances of detecting these genetic factors.

The concept for the Family Blood Pressure Program was conceived in the Report of the Expert Panel on Genetic Strategies for Heart, Lung, and Blood Diseases. The initiative was approved by the Arteriosclerosis, Hypertension, and Lipid Metabolism Advisory Committee (AHLMAC) in March, 1993. The genetic-epidemiological aspects were approved by the Clinical Applications and Prevention Advisory Committee (CAPAC) in February, 1993. The Request for Applications was released in March, 1994. Awards were made in September, 1995.

DESIGN NARRATIVE:

GENOA, the Genetic Epidemiology Network of Arteriopathy, consists of a network of three field centers and biochemical and genetic core labs to study the common polymorphic genetic variations to determine individual differences in blood pressure and essential hypertension in 1,500 sibling pairs in three racial groups. Linkage analyses are performed using an extensive array of candidate genes and anonymous markers throughout the genome.

Each collaborating investigator is responsible for an essential element of the network: Eric Boerwinkle for genotyping and linkage analyses, Robert Ferrell for genotyping, Craig Hanis for recruiting Mexican-Americans, Richard Hutchinson for recruiting African-Americans, Sharon Kardia for cladistic and prediction analyses and data management, and Stephen Turner for recruiting Non-Hispanic whites and measuring physiologic variables. Between 1995 and 2000, the network carried out five specific aims to localize and characterize the genetic determinants of high blood pressure. Aim 1 used robust sibling pair linkage methods in 500 hypertensive sibling pairs in each racial group (a total of 1,500 sibling pairs) to localize genes influencing interindividual differences in the occurrence of essential hypertension. Aims 2 and 3 took advantage of previously collected blood pressure and intermediate predictor trait data from 1,488 normotensive sibling pairs from the Rochester Family Heart Study to localize genes contributing to essential hypertension. The linkage analyses (Aims 1-3) used both an extensive array of candidate genes and a large number of anonymous markers throughout the genome. Aim 4 used multiple diallelic sequence polymorphisms and cladistic analyses within a linked gene to identify haplotypes for further DNA sequencing in order to identify candidate functional DNA sequence variation contributing to interindividual differences in BP levels and essential hypertension status. Aim 5 evaluated the ability of candidate functional DNA sequence variation to predict essential hypertension status in the three racial groups.

The study was renewed in September 2000 to pursue two lines of investigation. The first was to identify and characterize genes contributing to atherosclerotic coronary heart disease using electron beam computed tomography (EBCT) to quantify coronary artery calcification as a measure of preclinical disease. Robust sibling-pair linkage methods were used to determine whether any of the more than 375 highly polymorphic tandem repeat marker loci spanning the genome were linked to genes influencing EBCT measures of coronary artery calcification in at least 500 GENOA sibships from Rochester, Minnesota. Association analysis was used to determine whether biallelic markers of DNA sequence variation in candidate genes identified by GENOA or others to influence blood pressure level or diagnostic category also influence EBCT measures of coronary artery calcification in at least 500 GENOA participants from Rochester, Minnesota. The second line of investigation extended analytical methods (linkage disequilibrium regression and combinatorial partitioning) to more finely localize positional candidate genes and loci, and to identifying gene-gene and gene-environment interaction effects influencing the measured Family Blood Pressure Program and GENOA phenotypes.

In the next phase of the FBPP extending the study through FY 2008, a major emphasis is placed on making the Program a shared resource for hypertension researchers in the United States and throughout the world. In Aim 1, the intestigators will build, maintain and update a publicly available knowledge-base to facilitate research by non-FBPP investigators on the genetics of hypertension, its risk factors and its complications. In Aim 2, they will use state-of-the-art genetic linkage analysis methods to identify additional linkage regions using subgroups of pedigrees and physiologically relevant combinations of phenotypes that will aid in localizing hypertension genes. In Aim 3, they will use a combination of bioinformatics, a dense array of SNPs, and state-of-the-art data analysis to follow-up regions of interest and identify the underlying hypertension genes. The regions to be followed-up include those identified during the current phase of the FBPP and Aim 2 of this renewal phase. In Aim 4, they will evaluate the hypertension genes identified in Aim 3 for their association with multiple measures reflecting the cardiovascular and renal complications of hypertension, including left ventricular mass and microalbuminuria. It is the long-term goal of the FBPP to have the hypertension genetics community develop a comprehensive picture of the genetic architecture of human hypertension, including its risk factors, complications, and response to treatment.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Boerwinkle, Principal Investigator — University of Texas; Robert Ferrell, Principal Investigator — University of Pittsburgh; Craig Hanis, Principal Investigator — University of Texas; Sharon Kardia, Principal Investigator — University of Michigan; Thomas Mosley, Principal Investigator — University of Mississippi Medical Center; Stephen Turner, Principal Investigator — Mayo Clinic

REFERENCES:
- [Background] Boerwinkle E, Ellsworth DL, Hallman DM, Biddinger A. Genetic analysis of atherosclerosis: a research paradigm for the common chronic diseases. Hum Mol Genet. 1996;5 Spec No:1405-10. doi: 10.1093/hmg/5.supplement_1.1405. PMID 8875244
- [Background] Boerwinkle E. A contemporary research paradigm for the genetic analysis of a common chronic disease. Ann Med. 1996 Oct;28(5):451-7. doi: 10.3109/07853899608999107. PMID 8949978
- [Background] Page GP, Amos CI, Boerwinkle E. The quantitative LOD score: test statistic and sample size for exclusion and linkage of quantitative traits in human sibships. Am J Hum Genet. 1998 Apr;62(4):962-8. doi: 10.1086/301783. PMID 9529341
- [Background] Fornage M, Amos CI, Kardia S, Sing CF, Turner ST, Boerwinkle E. Variation in the region of the angiotensin-converting enzyme gene influences interindividual differences in blood pressure levels in young white males. Circulation. 1998 May 12;97(18):1773-9. doi: 10.1161/01.cir.97.18.1773. PMID 9603530
- [Background] Amos CI, Krushkal J, Thiel TJ, Young A, Zhu DK, Boerwinkle E, de Andrade M. Comparison of model-free linkage mapping strategies for the study of a complex trait. Genet Epidemiol. 1997;14(6):743-8. doi: 10.1002/(SICI)1098-2272(1997)14:63.0.CO;2-O. PMID 9433571
- [Background] Ellsworth DL, Hallman DM, Boerwinkle E. Impact of the Human Genome Project on epidemiologic research. Epidemiol Rev. 1997;19(1):3-13. doi: 10.1093/oxfordjournals.epirev.a017943. No abstract available. PMID 9360897
- [Background] Province MA, Boerwinkle E, Chakravarti A, Cooper R, Fornage M, Leppert M, Risch N, Ranade K. Lack of association of the angiotensinogen-6 polymorphism with blood pressure levels in the comprehensive NHLBI Family Blood Pressure Program. National Heart, Lung and Blood Institute. J Hypertens. 2000 Jul;18(7):867-76. doi: 10.1097/00004872-200018070-00008. PMID 10930184
- [Background] Bray MS, Li L, Turner ST, Kardia SL, Boerwinkle E. Association and linkage analysis of the alpha-adducin gene and blood pressure. Am J Hypertens. 2000 Jun;13(6 Pt 1):699-703. doi: 10.1016/s0895-7061(00)00242-9. PMID 10912756
- [Background] Boerwinkle E; Family Blood Pressure Program. All for one and one for all: introduction to a coordinated analysis of the Gly-460-Trp alpha-adducin polymorphism. Am J Hypertens. 2000 Jun;13(6 Pt 1):734-5. doi: 10.1016/s0895-7061(00)00243-0. No abstract available. PMID 10912761
- [Background] Bray MS, Krushkal J, Li L, Ferrell R, Kardia S, Sing CF, Turner ST, Boerwinkle E. Positional genomic analysis identifies the beta(2)-adrenergic receptor gene as a susceptibility locus for human hypertension. Circulation. 2000 Jun 27;101(25):2877-82. doi: 10.1161/01.cir.101.25.2877. PMID 10869257
- [Background] Krushkal J, Ferrell R, Mockrin SC, Turner ST, Sing CF, Boerwinkle E. Genome-wide linkage analyses of systolic blood pressure using highly discordant siblings. Circulation. 1999 Mar 23;99(11):1407-10. doi: 10.1161/01.cir.99.11.1407. PMID 10086961
- [Background] Turner ST, Boerwinkle E. Genetics of hypertension, target-organ complications, and response to therapy. Circulation. 2000 Nov 14;102(20 Suppl 4):IV40-5. doi: 10.1161/01.cir.102.suppl_4.iv-40. No abstract available. PMID 11080130
- [Background] Krushkal J, Xiong M, Ferrell R, Sing CF, Turner ST, Boerwinkle E. Linkage and association of adrenergic and dopamine receptor genes in the distal portion of the long arm of chromosome 5 with systolic blood pressure variation. Hum Mol Genet. 1998 Sep;7(9):1379-83. doi: 10.1093/hmg/7.9.1379. PMID 9700190
- [Background] Xiong MM, Krushkal J, Boerwinkle E. TDT statistics for mapping quantitative trait loci. Ann Hum Genet. 1998 Sep;62(Pt 5):431-52. doi: 10.1046/j.1469-1809.1998.6250431.x. PMID 10088040
- [Background] Bray MS, Boerwinkle E, Doris PA. High-throughput multiplex SNP genotyping with MALDI-TOF mass spectrometry: practice, problems and promise. Hum Mutat. 2001 Apr;17(4):296-304. doi: 10.1002/humu.27. PMID 11295828
- [Background] Wu X, Cooper RS, Borecki I, Hanis C, Bray M, Lewis CE, Zhu X, Kan D, Luke A, Curb D. A combined analysis of genomewide linkage scans for body mass index from the National Heart, Lung, and Blood Institute Family Blood Pressure Program. Am J Hum Genet. 2002 May;70(5):1247-56. doi: 10.1086/340362. Epub 2002 Mar 28. PMID 11923912
- [Background] Lange LA, Lange EM, Bielak LF, Langefeld CD, Kardia SL, Royston P, Turner ST, Sheedy PF 2nd, Boerwinkle E, Peyser PA. Autosomal genome-wide scan for coronary artery calcification loci in sibships at high risk for hypertension. Arterioscler Thromb Vasc Biol. 2002 Mar 1;22(3):418-23. doi: 10.1161/hq0302.105721. PMID 11884284
- [Background] Kardia SL, Rozek LS, Krushkal J, Ferrell RE, Turner ST, Hutchinson R, Brown A, Sing CF, Boerwinkle E. Genome-wide linkage analyses for hypertension genes in two ethnically and geographically diverse populations. Am J Hypertens. 2003 Feb;16(2):154-7. doi: 10.1016/s0895-7061(02)03249-1. PMID 12559685
- [Background] Province MA, Kardia SL, Ranade K, Rao DC, Thiel BA, Cooper RS, Risch N, Turner ST, Cox DR, Hunt SC, Weder AB, Boerwinkle E; National Heart, Lung and Blood Institute Family Blood Pressure Program. A meta-analysis of genome-wide linkage scans for hypertension: the National Heart, Lung and Blood Institute Family Blood Pressure Program. Am J Hypertens. 2003 Feb;16(2):144-7. doi: 10.1016/s0895-7061(02)03248-x. PMID 12559682
- [Background] Barkley RA, Brown AC, Hanis CL, Kardia SL, Turner ST, Boerwinkle E. Lack of genetic linkage evidence for a trans-acting factor having a large effect on plasma lipoprotein[a] levels in African Americans. J Lipid Res. 2003 Jul;44(7):1301-5. doi: 10.1194/jlr.M300163-JLR200. Epub 2003 May 1. PMID 12730294
- [Background] Morrison AC, Brown A, Kardia SL, Turner ST, Boerwinkle E; Genetic Epidemiology Network of Arteriopathy (GENOA) Study. Evaluating the context-dependent effect of family history of stroke in a genome scan for hypertension. Stroke. 2003 May;34(5):1170-5. doi: 10.1161/01.STR.0000068780.47411.16. Epub 2003 Apr 24. PMID 12714704
- [Background] Kullo IJ, McConnell JP, Bailey KR, Kardia SL, Bielak LF, Peyser PA, Sheedy PF 2nd, Boerwinkle E, Turner ST. Relation of C-reactive protein and fibrinogen to coronary artery calcium in subjects with systemic hypertension. Am J Cardiol. 2003 Jul 1;92(1):56-8. doi: 10.1016/s0002-9149(03)00466-1. No abstract available. PMID 12842247
- [Background] Turner ST, Jack CR, Fornage M, Mosley TH, Boerwinkle E, de Andrade M. Heritability of leukoaraiosis in hypertensive sibships. Hypertension. 2004 Feb;43(2):483-7. doi: 10.1161/01.HYP.0000112303.26158.92. Epub 2004 Jan 12. PMID 14718359
- [Background] Barkley RA, Chakravarti A, Cooper RS, Ellison RC, Hunt SC, Province MA, Turner ST, Weder AB, Boerwinkle E; Family Blood Pressure Program. Positional identification of hypertension susceptibility genes on chromosome 2. Hypertension. 2004 Feb;43(2):477-82. doi: 10.1161/01.HYP.0000111585.76299.f7. Epub 2004 Jan 19. PMID 14732741
- [Background] Daniels PR, Kardia SL, Hanis CL, Brown CA, Hutchinson R, Boerwinkle E, Turner ST; Genetic Epidemiology Network of Arteriopathy study. Familial aggregation of hypertension treatment and control in the Genetic Epidemiology Network of Arteriopathy (GENOA) study. Am J Med. 2004 May 15;116(10):676-81. doi: 10.1016/j.amjmed.2003.12.032. PMID 15121494
- [Background] O'Meara JG, Kardia SL, Armon JJ, Brown CA, Boerwinkle E, Turner ST. Ethnic and sex differences in the prevalence, treatment, and control of dyslipidemia among hypertensive adults in the GENOA study. Arch Intern Med. 2004 Jun 28;164(12):1313-8. doi: 10.1001/archinte.164.12.1313. PMID 15226165
- [Background] Morrison AC, Cooper R, Hunt S, Lewis CE, Luke A, Mosley TH, Boerwinkle E. Genome scan for hypertension in nonobese African Americans: the National Heart, Lung, and Blood Institute Family Blood Pressure Program. Am J Hypertens. 2004 Sep;17(9):834-8. doi: 10.1016/j.amjhyper.2004.04.009. PMID 15363828
- [Background] Kullo IJ, Bailey KR, Bielak LF, Sheedy PF 2nd, Klee GG, Kardia SL, Peyser PA, Boerwinkle E, Turner ST. Lack of association between lipoprotein(a) and coronary artery calcification in the Genetic Epidemiology Network of Arteriopathy (GENOA) study. Mayo Clin Proc. 2004 Oct;79(10):1258-63. doi: 10.4065/79.10.1258. PMID 15473406
- [Background] Kardia SL, Turner ST, Schwartz GL, Moore JH. Linear dynamic features of ambulatory blood pressure in a population-based study. Blood Press Monit. 2004 Oct;9(5):259-67. doi: 10.1097/00126097-200410000-00006. PMID 15472499
- [Background] Kullo IJ, Bailey KR, Kardia SL, Mosley TH Jr, Boerwinkle E, Turner ST. Ethnic differences in peripheral arterial disease in the NHLBI Genetic Epidemiology Network of Arteriopathy (GENOA) study. Vasc Med. 2003 Nov;8(4):237-42. doi: 10.1191/1358863x03vm511oa. PMID 15125483
- [Background] Frazier L, Turner ST, Schwartz GL, Chapman AB, Boerwinkle E. Multilocus effects of the renin-angiotensin-aldosterone system genes on blood pressure response to a thiazide diuretic. Pharmacogenomics J. 2004;4(1):17-23. doi: 10.1038/sj.tpj.6500215. PMID 14735111
- [Background] Tang H, Quertermous T, Rodriguez B, Kardia SL, Zhu X, Brown A, Pankow JS, Province MA, Hunt SC, Boerwinkle E, Schork NJ, Risch NJ. Genetic structure, self-identified race/ethnicity, and confounding in case-control association studies. Am J Hum Genet. 2005 Feb;76(2):268-75. doi: 10.1086/427888. Epub 2004 Dec 29. PMID 15625622
- [Background] Turner ST, Fornage M, Jack CR Jr, Mosley TH, Kardia SL, Boerwinkle E, de Andrade M. Genomic susceptibility loci for brain atrophy in hypertensive sibships from the GENOA study. Hypertension. 2005 Apr;45(4):793-8. doi: 10.1161/01.HYP.0000154685.54766.2d. Epub 2005 Feb 7. PMID 15699467
- [Background] An P, Freedman BI, Hanis CL, Chen YD, Weder AB, Schork NJ, Boerwinkle E, Province MA, Hsiung CA, Wu X, Quertermous T, Rao DC. Genome-wide linkage scans for fasting glucose, insulin, and insulin resistance in the National Heart, Lung, and Blood Institute Family Blood Pressure Program: evidence of linkages to chromosome 7q36 and 19q13 from meta-analysis. Diabetes. 2005 Mar;54(3):909-14. doi: 10.2337/diabetes.54.3.909. PMID 15734873
- [Background] Zhu X, Luke A, Cooper RS, Quertermous T, Hanis C, Mosley T, Gu CC, Tang H, Rao DC, Risch N, Weder A. Admixture mapping for hypertension loci with genome-scan markers. Nat Genet. 2005 Feb;37(2):177-81. doi: 10.1038/ng1510. Epub 2005 Jan 23. PMID 15665825
- [Background] Jorgenson E, Tang H, Gadde M, Province M, Leppert M, Kardia S, Schork N, Cooper R, Rao DC, Boerwinkle E, Risch N. Ethnicity and human genetic linkage maps. Am J Hum Genet. 2005 Feb;76(2):276-90. doi: 10.1086/427926. Epub 2004 Dec 30. PMID 15627237
- [Background] Klos KL, Kardia SL, Hixson JE, Turner ST, Hanis C, Boerwinkle E, Sing CF. Linkage analysis of plasma ApoE in three ethnic groups: multiple genes with context-dependent effects. Ann Hum Genet. 2005 Mar;69(Pt 2):157-67. doi: 10.1046/j.1529-8817.2004.00148.x. PMID 15720297
- [Background] Kraja AT, Rao DC, Weder AB, Mosley TH, Turner ST, Hsiung CA, Quertermous T, Cooper R, Curb JD, Province MA. An evaluation of the metabolic syndrome in a large multi-ethnic study: the Family Blood Pressure Program. Nutr Metab (Lond). 2005 Aug 2;2:17. doi: 10.1186/1743-7075-2-17. PMID 16076393
- [Background] Bielinski SJ, Lynch AI, Miller MB, Weder A, Cooper R, Oberman A, Chen YD, Turner ST, Fornage M, Province M, Arnett DK. Genome-wide linkage analysis for loci affecting pulse pressure: the Family Blood Pressure Program. Hypertension. 2005 Dec;46(6):1286-93. doi: 10.1161/01.HYP.0000191706.41980.29. Epub 2005 Nov 14. PMID 16286574
- [Background] Kullo IJ, Turner ST, Boerwinkle E, Kardia SL, de Andrade M. A novel quantitative trait locus on chromosome 1 with pleiotropic effects on HDL-cholesterol and LDL particle size in hypertensive sibships. Am J Hypertens. 2005 Aug;18(8):1084-90. doi: 10.1016/j.amjhyper.2005.02.010. PMID 16109322
- [Background] Levin AM, Ghosh D, Cho KR, Kardia SL. A model-based scan statistic for identifying extreme chromosomal regions of gene expression in human tumors. Bioinformatics. 2005 Jun 15;21(12):2867-74. doi: 10.1093/bioinformatics/bti417. Epub 2005 Apr 6. PMID 15814559
- [Derived] Scantlebury DC, Kane GC, Wiste HJ, Bailey KR, Turner ST, Arnett DK, Devereux RB, Mosley TH Jr, Hunt SC, Weder AB, Rodriguez B, Boerwinkle E, Weissgerber TL, Garovic VD. Left ventricular hypertrophy after hypertensive pregnancy disorders. Heart. 2015 Oct;101(19):1584-90. doi: 10.1136/heartjnl-2015-308098. Epub 2015 Aug 4. PMID 26243788